CLINICAL TRIAL: NCT07241494
Title: Investigation of Drug Use and Evaluation of Clinical Pharmacy Services in Patients With Renal Impairment.
Brief Title: Evaluation of Clinical Pharmacy Services and Drug Use in Renal Impairment.
Acronym: RECAP-Rx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Muhammed Yunus Bektay, Principle Investigator, Istanbul University - Cerrahpasa
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 18/12
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Renal Impairments; Chronic Kidney Disease; Acute Kidney Disease; Medication Errors
Keywords: Renal impairment; drug-related problems (DRPs); clinical pharmacist; pharmaceutical care; Clinical Pharmacy Services; Medication Errors; Chronic Kidney Disease; Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic; Renal Insufficiency; Kidney Diseases | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: This study uses a prospective, quasi-experimental design consisting of three consecutive patient groups: observation (control), education, and intervention. The groups were not randomised but were included sequentially over time in the same hospital setting. In the observation group, no clinical pharmacist intervention was provided. In the education group, physicians received structured training on renal dose adjustments for commonly prescribed medications. In the intervention group, the clinical pharmacist actively participated in daily ward rounds, identified and resolved drug-related problems (DRPs), and provided recommendations to physicians. Comparisons among the three groups were made to evaluate the effect of clinical pharmacy services and educational interventions on the identification and management of DRPs in patients with renal impairment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Observation Group (Control) (No Intervention): Patients with renal impairment hospitalised in the general internal medicine ward were monitored without any clinical pharmacist intervention. Prescriptions and drug use data were collected prospectively, and drug-related problems (DRPs) were identified retrospectively according to the Pharmaceutical Care Network Europe (PCNE) classification version 9.1. The results from this phase served as the baseline for comparison with subsequent groups.
- Education Group (Active Comparator): During this phase, physicians responsible for patient care received structured educational sessions delivered by the clinical pharmacist. The training focused on renal dose adjustment principles, identification of nephrotoxic drugs, and prevention of medication-related harm in patients with renal dysfunction. Patients admitted during this period were followed without direct pharmacist intervention. DRPs were identified and classified using the PCNE system to assess the indirect impact of education on prescribing behaviour.
  Interventions: Behavioral: Education for renal adjusments
- Intervention Group (Active Comparator): In this phase, the clinical pharmacist participated actively in daily ward rounds, performed comprehensive medication reviews, and identified drug-related problems (DRPs) using the Pharmaceutical Care Network Europe (PCNE) classification version 9.1. Interventions included recommendations for renal dose adjustments, correction of dosing errors, identification and prevention of drug-drug interactions, and optimisation of drug selection. The pharmacist communicated findings and recommendations directly to the treating physicians, and acceptance of interventions was documented.
  Interventions: Drug: Clinical Pharmacist-Led Pharmaceutical Care Service and Renal Dose Adjustment; Behavioral: Education for renal adjusments

INTERVENTIONS:
Drug: Clinical Pharmacist-Led Pharmaceutical Care Service and Renal Dose Adjustment — Clinical pharmacist-led interventions were implemented to optimise medication therapy and ensure patient safety among hospitalised patients with renal impairment. The interventions included several integrated pharmaceutical care activities conducted during daily ward rounds. The clinical pharmacist assessed renal function and adjusted medication doses according to up-to-date dosing guidelines and renal pharmacotherapy principles. In cases where inappropriate doses or dosing intervals were identified, corrective recommendations were communicated to the treating physicians to prevent under- or overdosing. The pharmacist also evaluated each patient's medication profile for potential drug-drug interactions and provided strategies to avoid clinically significant interactions. Drug selection was reviewed for indication, therapeutic appropriateness, and safety, with substitution or discontinuation proposed when necessary. In addition to these direct patient care activities, the clinical pharm
  Other Names: Renal Dose Adjustment; Drug-Drug Interaction Management; Correction of Dosing Errors; Optimisation of Drug Selection; Educational Feedback to Physicians
  Arms: Intervention Group
Behavioral: Education for renal adjusments — The educational intervention consisted of regular training sessions delivered by the clinical pharmacist to physicians on renal dose adjustment principles, identification of nephrotoxic drugs, and prevention of drug-related problems in patients with renal impairment. The sessions aimed to improve physicians' knowledge and prescribing practices for medications requiring renal dose modification.
  Arms: Education Group; Intervention Group

SUMMARY:
Clinical pharmacy services aim to optimise medication use, enhance patient outcomes, and reduce the risk of drug-related harm through patient-centred pharmaceutical care. In hospital settings, clinical pharmacists collaborate with physicians and other healthcare professionals as part of a multidisciplinary team to identify, prevent, and resolve drug-related problems (DRPs). Pharmacist interventions are defined as any action initiated by a pharmacist that directly contributes to patient management or results in a modification of medication therapy. The clinical and economic benefits of such interventions have been widely recognised in various healthcare environments.

This quasi-experimental study aims to investigate the impact of clinical pharmacy services on drug use and the management of DRPs in patients with renal impairment admitted to the general internal medicine ward. The study also evaluates the contribution of the clinical pharmacist to optimising the use of drugs that require renal dose adjustment.

The study was conducted in a university hospital and included three consecutive patient groups: observation (control), education, and intervention. In the observation group, no pharmacist intervention was performed. In the education group, physicians received a structured educational presentation on renal dose adjustment for commonly prescribed medications. In the intervention group, the clinical pharmacist actively participated in daily ward rounds, identified and resolved DRPs, and provided recommendations to physicians. DRPs were classified using the Pharmaceutical Care Network Europe (PCNE) classification version 9.1.

This study evaluates whether the integration of a clinical pharmacist into the healthcare team can improve the quality of pharmacotherapy, reduce DRPs-particularly those associated with renal dysfunction-and enhance patient safety and outcomes in hospitalised patients.

DETAILED DESCRIPTION:
Patients with renal impairment are at high risk for adverse drug reactions, medication errors, and inappropriate prescribing due to altered pharmacokinetics and pharmacodynamics. As renal function declines, dose adjustments and careful monitoring are required for many commonly prescribed drugs. Inappropriate dosing and the use of nephrotoxic agents in this population can lead to drug accumulation, toxicity, or therapeutic failure, thereby increasing the risk of hospitalisations, prolonged stays, and mortality. Previous studies have highlighted that a considerable proportion of drug-related hospital admissions are attributable to inadequate dose adjustment in patients with reduced kidney function. Therefore, careful monitoring and evidence-based dose optimisation are crucial in these patients.

Incorporating clinical pharmacy services into the care of patients with renal impairment may improve medication safety and treatment outcomes. Clinical pharmacists are well-positioned to identify and prevent drug-related problems (DRPs), recommend dose adjustments, and collaborate with physicians to enhance the quality of pharmacotherapy. Pharmacist-led interventions-such as medication reviews, dose optimisation, education of healthcare providers, and direct communication of recommendations-have been shown to reduce medication errors and improve patient outcomes in various clinical settings. Furthermore, integrating clinical pharmacists into multidisciplinary hospital teams has demonstrated positive impacts on treatment effectiveness, patient safety, and overall healthcare costs.

The present study aims to investigate drug use patterns, identify DRPs, and evaluate the impact of clinical pharmacy services on the management of patients with renal impairment admitted to the general internal medicine ward. The study specifically focuses on the pharmacist's role in optimising drug therapy for medications requiring renal dose adjustments. By assessing both the educational and interventional contributions of clinical pharmacists, this study intends to provide evidence supporting the integration of these services into routine hospital practice.

This study adopts a prospective, quasi-experimental design and was conducted in the general internal medicine ward of a university hospital. Three consecutive patient groups were included: the observation (control) group, the education group, and the intervention group. In the observation group, patients were followed without any direct pharmacist intervention. In the education group, physicians received structured training on renal dose adjustment principles and the safe use of frequently prescribed medications in renal dysfunction. In the intervention group, the clinical pharmacist actively participated in daily ward rounds, performed comprehensive medication reviews, and identified DRPs related to inappropriate drug selection, dosage errors, potential drug-drug interactions, and drugs requiring renal adjustment. The clinical pharmacist provided evidence-based recommendations to physicians regarding clinically significant findings, and these interventions were documented systematically.

All identified DRPs were classified according to the Pharmaceutical Care Network Europe (PCNE) classification system version 9.1. The clinical pharmacist's recommendations and physician acceptance rates were also recorded. Patient data-including demographic information, comorbidities, renal function parameters, prescribed medications, and relevant laboratory results-were collected prospectively. Statistical comparisons were made between the three study groups to evaluate the effect of educational and interventional phases on the frequency and nature of DRPs, particularly those associated with renal dysfunction.

Through this design, the study aims to demonstrate the stepwise impact of clinical pharmacy involvement-from passive observation to educational and active interventional roles-on the rational use of medicines in patients with renal impairment. It is expected that increased clinical pharmacist participation will lead to a reduction in DRPs, particularly those related to renal dosing errors, and improve patient outcomes by ensuring safer and more effective medication use. The findings are anticipated to contribute to the development of standardised clinical pharmacy service models and support the integration of pharmacists into multidisciplinary care teams for patients with chronic kidney disease and related comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalised in the General Internal Medicine ward with an estimated glomerular filtration rate (eGFR) below 60 mL/min/1.73 m².
* Hospital stay of at least 48 hours.
* Receiving at least one medication that requires dose adjustment in renal impairment.
* Age 18 years or older.

Exclusion Criteria:

* eGFR value of 60 mL/min/1.73 m² or higher.
* Not receiving any medication that requires renal dose adjustment.
* Hospital stay shorter than 48 hours.
* Age under 18 years.
* Refusal or inability to provide informed consent.
* Lack of sufficient cognitive ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-10-31 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Change in the number of drug-related problems (DRPs) per patient | 12 months
  The total number of drug-related problems (DRPs) identified per patient, classified according to the Pharmaceutical Care Network Europe (PCNE) Classification System Version 9.1. This outcome measures the effect of clinical pharmacist-led educational and interventional activities on the identification and management of DRPs, with a specific focus on those associated with renal dysfunction.

SECONDARY OUTCOMES:
Percentage of drug-related problems (DRPs) associated with renal dysfunction | 12 months
  The percentage of total drug-related problems (DRPs) that are directly associated with renal dysfunction, including inappropriate drug selection, dosing errors, or the use of contraindicated medications. This outcome assesses the impact of clinical pharmacist-led educational and interventional activities on improving renal dose adjustment practices.
Acceptance rate of pharmacist recommendations by physicians | 12 months
  The proportion of pharmacist interventions or recommendations accepted and implemented by physicians in the intervention phase. This measure assesses the feasibility, acceptance, and clinical relevance of clinical pharmacist contributions to the multidisciplinary care team.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed Yunus BEKTAY, PHD, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared due to ethical necessities.